CLINICAL TRIAL: NCT04506931
Title: Comparison of Short Message Service (SMS), Interactive Voice Response (IVR), and Computer Assisted Telephone Interview (CATI) Mobile Phone Surveys for Non-communicable Disease Risk Factor Surveillance in Colombia
Brief Title: Comparison of SMS, IVR, and CATI Surveys in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318 - xyz
Record Dates: First submitted 2020-08-07; First posted 2020-08-10 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; computer assisted telephone interview; short message service; non-communicable diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of three mobile phone survey modalities: 1) SMS; 2) IVR; 3) CATI.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short Message Service (SMS) survey (Experimental): Participants will receive an SMS survey
  Interventions: Other: SMS Survey
- Interactive Voice Response (IVR) survey (Experimental): Participants will receive an IVR survey
  Interventions: Other: IVR Survey
- Computer Assisted Telephone Interviews (CATI) survey (Experimental): Participants will receive a CATI survey
  Interventions: Other: CATI Survey

INTERVENTIONS:
Other: SMS Survey — Participants will receive a SMS survey
  Arms: Short Message Service (SMS) survey
Other: IVR Survey — Participants will receive an IVR survey
  Arms: Interactive Voice Response (IVR) survey
Other: CATI Survey — Participants will receive a CATI survey
  Arms: Computer Assisted Telephone Interviews (CATI) survey

SUMMARY:
The objective of the study is to adapt and assess the feasibility, quality, and validity of short message service or 'text message' (SMS), interactive voice response (IVR), and computer assisted telephone interviews (CATI) for collecting information on noncommunicable disease (NCD) risk factors

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling technique, RDD participants will be randomized to one of the three arms: 1) SMS or 2) IVR or 3) CATI. Participants in the first study arm will receive an SMS survey. Participants in the second study arm will receive a IVR survey. Participants in the third study arm will receive a CATI survey. The IVR, SMS and CATI questionnaires contain a set of demographic questions and one NCD module (alcohol, or tobacco, or diet, or physical activity, or blood pressure and diabetes). The investigators will examine contact, response, refusal and cooperation rates and demographic representativeness by each study arm.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Colombia, conversant in the Spanish language

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5676 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is the number of participants with complete interviews, P is the number of participants with partial interviews, and R is the number of participants with refusals and breakoffs.
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is the number of participants with complete interviews, P is the number of participants with partial interviews, R is the number of participants with refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is the number of participants with refusals and breakoffs, I is the number of participants with complete interviews, P is the number of participants with partial interviews, and eU is the estimated eligible proportion of unknowns
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is the number of participants with complete interviews, P is the number of participants with partial interviews, R is the number of participants with refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Gibson, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; Angelica T Quinterro, PhD, MD, MSc, Principal Investigator — Pontificia Universidad Javeriana
Locations (1):
- Pontificia Universidad Javeriana, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722